CLINICAL TRIAL: NCT04850716
Title: An Observational Study of Relationship Between Standard Treatment Efficacy and The Tumor Microenvironment in Advanced Gastric Cancer
Brief Title: Relationship Between Standard Treatment Efficacy and The Tumor Microenvironment in Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2019-264
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Tumor Microenvironment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
Gastric cancer is among the most common malignant tumors nationwide with high morbidity and mortality. Attributing to its insidious onset and rapid progress, 70% of patients with gastric cancer were initially diagnosed at an advanced stage. In advanced gastric cancer, systemic treatment based on chemotherapy drugs, targeted drugs, and immune checkpoint inhibitors remains the main regimens. Among current standard treatment regimens, though HER2-positive and MSI-H/dMMR statuses indicate the treatment efficacy of trastuzumab and immune checkpoint inhibitors, there is still lack of robust biomarkers for predicting treatment efficacy. Tumor microenvironment as pivotal components of solid tumor, significantly influences therapeutic response and clinical outcome. The study is a multi-center, observational study to evaluate the relationship between standard treatment efficacy and the tumor microenvironment in advanced gastric cancer. In addition, the study comprehensively evaluated the landscape of the tumor microenvironment characteristics of gastric cancer, and aimed at establishing robust biomarkers for predicting prognosis and treatment efficacy to finetune treatment strategies.

DETAILED DESCRIPTION:
Gastric cancer is among the most common malignant tumors nationwide with high morbidity and mortality. Attributing to its insidious onset and rapid progress, 70% of patients with gastric cancer were initially diagnosed at an advanced stage. In advanced gastric cancer, systemic treatment based on chemotherapy drugs, targeted drugs, and immune checkpoint inhibitors remains the main regimens. Among current standard treatment regimens, though HER2-positive and MSI-H/dMMR statuses indicate the treatment efficacy of trastuzumab and immune checkpoint inhibitors, there is still lack of robust biomarkers for predicting treatment efficacy. Tumor microenvironment as pivotal components of solid tumor, significantly influences therapeutic response and clinical outcome. The study is a multi-center, observational study to evaluate the relationship between standard treatment efficacy and the tumor microenvironment in advanced gastric cancer. In addition, the study comprehensively evaluated the landscape of the tumor microenvironment characteristics of gastric cancer, and aimed at establishing robust biomarkers for predicting prognosis and treatment efficacy to finetune treatment strategies. Eligible subjects were selected according to the inclusion criteria and exclusion criteria. After successful screening, the patients were treated following the clinical guidelines and the actual conditions. The residual tissue samples of the primary tumor or metastatic foci were collected to conduct the tumor microenvironment detection analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced gastric cancer.
2. Willing to receive anti-tumor drug treatment.
3. Willing to provide residual tumor tissues after routine clinical diagnosis for tumor microenvironment detection analysis.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
5. At least one measurable lesion or non-measurable but evaluable as defined by RECIST 1.1.

Exclusion Criteria:

1. Human epidermal growth factor receptor 2 (HER2) is positive, that is, tissue immunohistochemical staining (IHC) (3+) or IHC (2+), and tissue fluorescence in situ hybridization (FISH) is positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed advanced gastric cancer.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 4 years
  Defined as the time from initiation date of first cycle to the first documentation of disease progression by independent review or to death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 4 years
  Defined as the percentage of patients who had a best response of complete response (CR), or partial response (PR).
Overall Survival (OS) | 4 years
  Defined as the time from initiation date of first cycle until the date of first documented date of death from any cause.
Duration Of Response (DOR) | 4 years
  Defined as the time from first documented response to first documented tumor progression or death from any cause.
Disease Control Rate (DCR) | 4 years
  Defined as the percentage of patients who had a best response of complete response (CR), partial response (PR), or stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No